CLINICAL TRIAL: NCT02555670
Title: Relation Between Bioelectrical Impedance-derived Muscle Mass and CT-derived Muscle Area in Critically Ill Patients
Brief Title: Relation Between Bioelectrical Impedance Analysis (BIA) and CT-scan Analysis in the ICU
Acronym: ICUBIACT
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Wilhelmus G.P.M. Looijaard, MD, PhD Candidate, Amsterdam UMC, location VUmc
Other Study IDs: ICUBIACT
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Muscular Atrophy
Keywords: Muscles; Intensive Care; Tomography, X-Ray Computed; Electric Impedance
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BIA and CT: Patients who had a CT-scan made for diagnostic reasons.
  Interventions: Other: BIA

INTERVENTIONS:
Other: BIA — Bioelectrical impedance analysis was performed within 4 days after a CT-scan was made
  Other Names: Bioelectrical impedance analysis

SUMMARY:
Aim of the present study is to determine whether muscle mass as assessed by bioelectrical impedance analysis correlates with and corresponds to muscle mass as assessed by CT scan analysis in critically patients admitted to the intensive care unit.

DETAILED DESCRIPTION:
BIA measurements are performed in critically ill patients admitted to the ICU or MC, within 72 hours before or after CT scanning.

The BIA measurements are taken with the BIA 101 ASE, manufactured by Akern, Florence-7 Italy. This device is phase sensitive and injects an alternating current of 400 µA at 50 kHz. Measurements were performed while patients lay in supine position with a pillow supporting the head. The resistance, reactance, body weight and length are entered in the BIA algorithm, using BodyGram PRO. This algorithm calculated the body composition, with muscle mass being reported in kilogram (kg).

Abdominal CT scans are analyzed using the computer program SliceOmatic® version 4.3 and 5.0 (TomoVision, Montreal, QC, Canada) at the level of the third lumbar vertebra (L3). The muscle tissue was identified by using boundaries in Hounsfield Units (grayscale) set of -29 to +150(23). The program computes muscle surface area in cm2, by multiplying the pixel area by the amount of pixels identified as muscle.

For a direct comparison with the BIA-derived muscle mass, the CT-derived muscle area is converted to kg. This is done by following two steps. Firstly, the Shen equation is used for the conversion to litres.Secondly, the muscle volume is multiplied by its density, resulting in muscle mass expressed in kg.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal CT-scan made for diagnostic reasons

Exclusion Criteria:

* CT-scan not analysable
* Internal or external metal devices
* active pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Adult Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Agreement between BIA-derived muscle mass and CT-derived muscle mass | Patient's data from the ICU-stay will be used, an average of one week
  Agreement will be calculated using a Bland-Altman plot

SECONDARY OUTCOMES:
Sensitivity of BIA to identify low muscle patients | Patient's data from the ICU-stay will be used, an average of one week
  Using CT-derived cut-off points, sensitivity of BIA to identify the same patients as having low muscle will be calculated
Specificity of BIA to identify low muscle patients | Patient's data from the ICU-stay will be used, an average of one week
  Using CT-derived cut-off points, specificity of BIA to identify the same patients as having low muscle will be calculated
Correlation between BIA-derived muscle mass and CT-derived muscle mass | Patient's data from the ICU-stay will be used, an average of one week
  Correlation will be calculated using Pearson's r

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelmus Looijaard, MD, Principal Investigator — Amsterdam UMC, location VUmc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weijs PJ, Looijaard WG, Dekker IM, Stapel SN, Girbes AR, Oudemans-van Straaten HM, Beishuizen A. Low skeletal muscle area is a risk factor for mortality in mechanically ventilated critically ill patients. Crit Care. 2014 Jan 13;18(2):R12. doi: 10.1186/cc13189. PMID 24410863
- [Derived] Looijaard WGPM, Stapel SN, Dekker IM, Rusticus H, Remmelzwaal S, Girbes ARJ, Weijs PJM, Oudemans-van Straaten HM. Identifying critically ill patients with low muscle mass: Agreement between bioelectrical impedance analysis and computed tomography. Clin Nutr. 2020 Jun;39(6):1809-1817. doi: 10.1016/j.clnu.2019.07.020. Epub 2019 Aug 10. PMID 31492456